CLINICAL TRIAL: NCT01104844
Title: Multicentre, Double-blind, Placebo-controlled, Randomized, Parallel Group Comparison of the Analgesic Effects of Different Maxigesic Doses Versus Acetaminophen, Ibuprofen and Placebo for the Teeth Extraction Pain
Brief Title: Maxi-Analgesic Phase 2 Study to Compare the Analgesic Effects in Different Dosing Groups to Treat Teeth Extraction Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn due to administrative reason
Sponsor: AFT Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFT-MX-3
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Dental Pain
Keywords: dental pain; Analgesia
MeSH Terms: conditions — Toothache; Agnosia | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Half dose strength (Active Comparator): Investigational drug half dose strength (acetaminophen 250mg + ibuprofen 75mg), i.e 2 tablets equating to ½ the dose in the standard investigational drug
  Interventions: Drug: Half dose strength
- Quarter dose strength (Active Comparator): Investigational drug quarter dose strength (acetaminophen125mg + Ibuprofen 37.5mg) i.e. 2 tablets equating to ¼ the dose in the standard investigational drug.
  Interventions: Drug: Quarter dose strength
- Acetaminophen standard dose (Active Comparator): Acetaminophen standard dose 500mg i.e. 2 tablets equating to the same acetaminophen dose as in the standard investigational drug
  Interventions: Drug: Acetaminophen standard dose
- ibuprofen low dose (Active Comparator): Ibuprofen low dose 150mg tablet i.e. 2 tablets equating to the same ibuprofen dose as in the standard investigational product
  Interventions: Drug: Ibuprofen low dose
- Ibuprofen high dose (Active Comparator): Ibuprofen High dose 300mg i.e. 2 tablets equating to twice the ibuprofen dose as in the standard investigational drug
  Interventions: Drug: Ibuprofen high dose
- placebo (Placebo Comparator): 2 Placebo tablets
  Interventions: Drug: Placebo
- Full Dose Strength (Experimental): Investigational drug full dose strength (acetaminophen 500mg + ibuprofen 150mg) i.e. 2 tablets
  Interventions: Drug: Full Dose Strength

INTERVENTIONS:
Drug: Full Dose Strength — Acetaminophen + ibuprofen, 2 tablets every 6 hours, with food for 24 hours (i.e a total of 4 x 1000/300 mg doses of study drug comprising of 8 tablets)
  Other Names: Brand name Maxigesic
  Arms: Full Dose Strength
Drug: Quarter dose strength — Investigational drug quarter dose strength (acetaminophen 125mg + ibuprofen 37.5mg) i.e. 2 tablets equating to 1/4 the dose in the standard investigational drug.
  Other Names: Maxigesic Quarter Dose
  Arms: Quarter dose strength
Drug: Half dose strength — Investigational drug half dose strength (acetaminophen 250mg + ibuprofen 75mg) i.e. 2 tablets equating to 1/2 the dose in the standard investigational drug
  Other Names: Maxigesic half dose
  Arms: Half dose strength
Drug: Acetaminophen standard dose — Acetaminophen standard dose 500mg i.e. 2 tablets equating to the same acetaminophen dose as in the standard investigational drug
  Other Names: paracetamol
  Arms: Acetaminophen standard dose
Drug: Ibuprofen low dose — Ibuprofen low dose 150mg tablet i.e. 2 tablets equating to the same ibuprofen dose as in the standard investigational product
  Other Names: Ibuprofen
  Arms: ibuprofen low dose
Drug: Ibuprofen high dose — Ibuprofen high dose 300mg i.e. 2 tablet equating to twice the ibuprofen dose as in the standard investigational drug
  Other Names: Ibuprofen
  Arms: Ibuprofen high dose
Drug: Placebo — 2 placebo tablets
  Arms: placebo

SUMMARY:
The aim of the study is to examine the dose response relationship in the treatment of dental pain (teeth extraction) for the different potential doses of the investigational drug, i.e. 2 tablets, 1 tablet or ½ a tablet given 4 times a day.

DETAILED DESCRIPTION:
The combination of 500 mg acetaminophen and 150 mg ibuprofen has been shown to improve analgesia compared with the individual components, when given as 2 tablets (i.e., total of 1,000/300 mg) 4 times a day for dental pain.

The analgesic relief from 2 tablets of the combination was around 6 hours, and so consistent with 4 times a day dosing.

The combination tablets are scored to allow for lower doses and can be given as 2 tablets (total of 1,000/300 mg), 1 tablet (500/150 mg) or ½ tablet (250/75 mg) in multiple doses.

However different dose response combinations need to be investigated to confirm the dose response curve of the combination and to compare the relative efficacy with acetaminophen and different doses of ibuprofen (lower and higher dose).

The study hypothesis is the analgesic response to three different combination doses, the three single component doses 500mg acetaminophen and 150mg and 300mg ibuprofen, and placebo administered four times daily over 24 hours for post-operative dental pain will form a representative dose response curve.

The study design is multi-centre, prospective, placebo-controlled, randomized, double-blind, factorial parallel group.

Participants will be stratified for baseline pain at inclusion (moderate or severe pain based a 4 point pain intensity rating scale).

Recruitment will continue until there are at least 350 participants in the ITT population.

Efficacy: The primary efficacy objective is to compare the time-adjusted SPIDs (Summed Pain Intensity Differences) of the VAS pain intensity scores up to 24 hours after the first dose of study medication among the 7 treatment groups to determine the form of the dose-response relationship.

Secondary efficacy objectives are:

* To compare the maximum VAS pain scores for the 24-hour period after the first dose of study medication among the seven treatment groups to determine the form of the dose response relationship.
* To compare the response rates (response rate to be defined as the percentage of participants who achieve at least 50% reduction in baseline pain within 6 hours i.e. the first dose period) among the seven treatment groups to determine the form of the dose response relationship.
* To determine and compare the time to peak reduction in VAS pain intensity scores following the first dose of study medication among the seven treatment groups to determine the form of the dose response relationship.
* To compare time to perceptible and meaningful pain relief among the seven treatment groups using the two stopwatch method.
* To compare the time to requirement for rescue medication among the seven treatment groups.
* To compare the amount of rescue medication used (defined as the number of tablets) among the seven treatment groups over the 24-hour treatment period.
* To compare the percentage of participants requiring rescue medication among the seven treatment groups.
* To compare the categorical global pain rating among the seven treatment groups.

Safety:

To compare adverse event rates (divided into serious and non-serious adverse events). Adverse events will be assessed for the 24- hour study period and up to 30 days after the final dose of study medication among the seven treatment groups.

The standard symptoms expected in subjects who have recently undergone third molar extraction will not be recorded as AEs in this study, unless they are of greater severity and/or intensity than would be expected. The events considered to be standard for the purposes of this study are:

* Oral pain.
* Facial swelling.
* Oral bleeding.
* Bruising to face, neck, and/or jaw.
* Decreased range of motion of the jaw.
* Dry socket.

The Investigators will use their clinical judgement in determining whether these symptoms are of greater severity and/or intensity than would be expected.

Planned hospital admissions and/or surgical operations for an illness or disease which existed before the drug was given or the participant was randomized in a clinical study will not be considered adverse events The incidence of known specific NSAID and acetaminophen side effects (e.g. GI ulceration, Indigestion/stomach pain, post-operative bleeding, thromboembolic events and evidence of clinical hepatitis) during the 24-hour study period and up to 30 days after the last dose will be compared among the seven treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before initiation of any study-related procedures.
2. Males and females aged at least 16 years and not more than 40 years old on the day of consent.
3. Undergoing oral surgery for the extraction of 2 impacted 3rd molar teeth, one of which must be mandibular and require bone removal.
4. Experiencing moderate to severe post-operative pain, as defined by a 4 point categorical pain intensity rating scale with 0 = no pain; 1 = mild pain; 2 = moderate pain and 3 = severe pain(at rest) within 6 hours after completion of surgery.
5. Baseline VAS pain intensity score of > 50mm on a 100mm VAS scale with 0 = no pain and 100 = worst pain imaginable.

Exclusion Criteria:

Study contra-indications:

1. Has taken any NSAID or acetaminophen within 12 hours prior to the start of surgery other than aspirin ≤ 150mg/day.
2. Subjects who have received any anesthetics from midnight the night prior to surgery, except for lidocaine with epinephrine, nitrous oxide, diazepam (Valium®), methohexital (Brevital®).
3. Known to be pregnant or possibly pregnant.
4. Women of childbearing potential who are unwilling to take adequate contraceptive precautions, i.e., a hormonal contraceptive, an intrauterine device, double-barrier method, or abstinence (should the subject become sexually active, she must agree to use a double-barrier method of contraception). A woman of childbearing potential is defined as any female who is less than 2 years post-menopausal or has not undergone a partial or total hysterectomy or surgical sterilization, e.g., bilateral tubal ligation, bilateral oophorectomy.
5. Suffering from a neurological disorder relating to pain perception or any acute or chronic condition that, in the opinion of the investigator, makes the subject unsuitable from an efficacy or safety perspective.
6. In the opinion of the investigator, unable to understand the visual analogue pain score or comply with the protocol requirements.
7. Currently or in last 30 days, has been in a clinical trial involving another study drug.
8. Currently treated with an ACE inhibitor, warfarin, steroid (other than nasal steroids or topical steroids with the approval of the investigator), cyclosporin, tacrolimus or methotrexate, or any other medication felt by the investigator to interfere with safety or efficacy evaluations.
9. Participant weight < 50kg.Suffering from any other diseases or condition which, in the opinion of the investigator, means that it would not be in the participant's best interests to participate in this study.

   NSAID and/or acetaminophen contra-indications:
10. Hypersensitivity to aspirin or other NSAID.
11. Hypersensitivity to acetaminophen.
12. Severe known hemopoietic, renal or hepatic disease, or immunosuppressed.
13. History of gastric ulceration or other GI disorders that, in the opinion of the investigator make the subject unsuitable (e.g., frequent treatment of GERD, inflammatory bowel disease, etc.).
14. History of severe asthma defined as asthma requiring frequent or ongoing treatment to control symptoms. Exercise-induced asthma or mild asthma not requiring ongoing treatment may not be exclusionary at the discretion of the investigator.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
the time-adjusted SPIDs of the VAS pain intensity scores | 24 hours after the first dose
  The primary efficacy objective is to compare the time-adjusted SPIDs of the VAS pain intensity scores up to 24 hours after the first dose of study medication among the 7 treatment groups to determine the form of the dose-response relationship.

SECONDARY OUTCOMES:
the maximum VAS pain score | 24 hours after the first dose
  To compare the maximum VAS pain scores for the 24-hour period after the first dose of study medication among the seven treatment groups to determine the form of the dose response relationship.
The Response Rate | 24 hours after the first dose
  To compare the response rates (response rate to be defined as the percentage of participants who achieve at least 50% reduction in baseline pain within 6 hours i.e. the first dose period) among the seven treatment groups to determine the form of the dose response relationship.
The time to peak reduction in VAS pain intensity scores | 24 hours after the first dose
  To determine and compare the time to peak reduction in VAS pain intensity scores following the first dose of study medication among the seven treatment groups to determine the form of the dose response relationship.
The time to perceptible and meaningful pain relief | 24 hours after the first dose
  To compare time to perceptible and meaningful pain relief among the seven treatment groups using the two stopwatch method.
The time to requirement for rescue medication | 24 hours after the first dose
  To compare the time to requirement for rescue medication among the seven treatment groups.
The amount of rescue medication used | 24 hours after the first dose
  To compare the amount of rescue medication used (defined as the number of tablets) among the seven treatment groups over the 24-hour treatment period.
The percentage of participants requiring rescue medication | 24 hours after the first dose
  To compare the percentage of participants requiring rescue medication among the seven treatment groups.
The categorical global pain rating | 24 hours after the first dose
  To compare the categorical global pain rating among the seven treatment groups which is obtained at the end of 24 hours study period.
The incidence of adverse events | up to 30 days after the last dose
  Adverse events (divided into serious and non-serious adverse events) will be assessed for the study period. Adverse events will also be determined up to 30 days after the last dose.
  The incidence of individual specific NSAID and acetaminophen side effects (e.g. GI ulceration, indigestion/stomach pain, post-operative bleeding and evidence of clinical hepatitis) will be determined up to 30 days after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuss, Doctor, Principal Investigator — Premier Research Group Ltd.
Locations (1):
- Austin Clinic, Austin, Texas, United States

REFERENCES:
- [Background] Merry AF, Gibbs RD, Edwards J, Ting GS, Frampton C, Davies E, Anderson BJ. Combined acetaminophen and ibuprofen for pain relief after oral surgery in adults: a randomized controlled trial. Br J Anaesth. 2010 Jan;104(1):80-8. doi: 10.1093/bja/aep338. PMID 20007794
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348